CLINICAL TRIAL: NCT02264262
Title: Noninvasive Measurement of Sympathetic Nerve Activity in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PRO00036916
Record Dates: First submitted 2014-10-07; First posted 2014-10-15 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2017-08

CONDITIONS: Sympathetic Nerve Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sympathetic nerve activity (Experimental): Healthy volunteers will undergo microneurography, and non invasive sympathetic nerve activity by EKG analysis at baseline and in response to stress.
  Interventions: Other: Physiologic maneuvers

INTERVENTIONS:
Other: Physiologic maneuvers — Subjects will perform cold pressor test, valsalva maneuver, hand grip and post-exercise occlusion in a controlled research environment

SUMMARY:
Activation of the sympathetic nervous system is associated with increased risk of ventricular arrhythmias and sudden cardiac death (SCD). Development of simple, noninvasive, reliable tools to measure sympathetic outflow in human subjects is therefore highly desirable.

Microneurography is the current gold standard measurement technique, whereby multiunit postganglionic sympathetic nerve activity is recorded with tungsten ultrafine microelectrodes inserted selectively into nerve fascicles of the peroneal nerve. Though this technique is considered extremely safe, and has been used successfully for decades in human translational physiology experiments, it has not been adopted for routine clinical assessment due to the requirement for sophisticated equipment and specific technical training and skills. Alternatively, many have adopted heart rate variability as a simple, noninvasive technique for assessing sympathetic nerve activity. However, heart rate variability does not directly measure sympathetic nerve activity, and there is much debate in the literature as to the exact source of sympathetic nerve traffic. For example, many believe it is an accurate reflection of cardiac sympathetic nerve activity, but does not accurately reflect changes in muscle or skin sympathetic nerve activity.

To address these limitations, the investigators have developed a simple, noninvasive technique to measure sympathetic nerve activity using surface electrodes.

Despite its great promise, this new approach has not yet been directly validated. The purpose of this study is therefore to validate this new technique (refered to as EKG-NA) against the current gold standard measurement technique, microneurography.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years of age
* BMI < 35 kg/m2

Exclusion Criteria:

* History of hypertension, diabetes, pulmonary disease, metabolic disease or heart failure
* Cardiac rhythm disorder, specifically: rhythm other than sinus
* Use of any medications other than common supplements
* Unable to perform handgrip exercise
* Pregnant

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2014-10; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Chane in Sympathetic nerve activity | Change from baseline in sympathetic nerve activity at 2 hours
  Multi-unit recordings of sympathetic nerve activity will be obtained with single-use sterile tungsten microelectrodes inserted selectively into muscle or skin nerve fascicles of the peritoneal nerve and EKG-NA by standard surface electrodes

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Victor, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States